CLINICAL TRIAL: NCT06531668
Title: A Clinical Trial to Examine the Efficacy of a Supplement to Support Hormone Regulation in Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scale Media Inc (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20431
Record Dates: First submitted 2024-07-17; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Hormone Regulation
Keywords: Women's Health; Menstrual Cycle; Estrogen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beyond Hormone Supplement (Experimental): Participants in this arm will receive the Beyond Hormone supplement.
  Interventions: Dietary Supplement: Beyond Hormone
- Placebo (Placebo Comparator): Participants in this arm will receive a placebo consisting of rice flour encapsulated in a vegetable cellulose capsule.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Beyond Hormone — Participants will take three capsules once daily with their morning meal for the duration of three menstrual cycles.
  Arms: Beyond Hormone Supplement
Other: Placebo — Participants will take three capsules once daily with their morning meal for the duration of three menstrual cycles.
  Arms: Placebo

SUMMARY:
This randomized, triple-blind, placebo-controlled trial will evaluate the efficacy of Live Conscious's Beyond Hormone supplement in regulating hormone production in women. The study involves 50 generally healthy female participants aged 25-45 who are not menopausal. The trial spans three menstrual cycles and assesses both objective hormone levels and subjective well-being through blood tests and questionnaires, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Female at-birth, aged 25-45.
* Not menopausal or perimenopausal.
* Regularly menstruating.
* Not taking any medication, supplement, or vitamin affecting hormone levels.
* Generally healthy and not living with any uncontrolled chronic disease.

Exclusion Criteria:

* Medical conditions or treatments affecting hormonal regulation.
* Endocrine disorders, gynecological or reproductive health conditions.
* Use of hormonal contraceptives or hormone therapy.
* Recent major illness or surgery.
* Severe allergies or hypersensitivities.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2024-09-07 (Estimated); Study Completion 2024-09-07 (Estimated)

PRIMARY OUTCOMES:
Hormone Levels Blood Panel (estradiol, testosterone, DHEA, insulin, and progesterone) | Baseline (Day 0), Midline (Day 45), and Endline (Day 90)
  Measurement of hormone levels. Blood tests will be conducted to evaluate these levels at Baseline (Day 2-5 of the first menstrual period), Midline (Day 2-5 of the second menstrual period), and Endline (Day 2-5 of the third menstrual period).

SECONDARY OUTCOMES:
Participants' Perceptions of Quality of Life | Baseline (Day 0), Midline (Day 45), and Endline (Day 90)
  Evaluation of participants' perceptions of the product's effects on quality of life with a self-reported questionnaire.
Participants' Mood and Energy Levels using the Visual Analog Scale (VAS) | Baseline (Day 0), Midline (Day 45), and Endline (Day 90)
  Assessment of participants' mood and energy levels using the Visual Analog Scale (VAS). These assessments will be conducted at Baseline (Day 2-5 of the first menstrual period), Midline (Day 2-5 of the second menstrual period), and Endline (Day 2-5 of the third menstrual period).
Participants' Monthly Cycle Symptoms using the Menstrual Cycle Symptom Diary (MCSD) | Baseline (Day 0), Midline (Day 45), and Endline (Day 90)
  Evaluation of participants' monthly cycle symptoms using the Menstrual Cycle Symptom Diary (MCSD). These assessments will be conducted at Baseline (Day 2-5 of the first menstrual period), Midline (Day 2-5 of the second menstrual period), and Endline (Day 2-5 of the third menstrual period).
Participants' Libido using a Libido Questionnaire | Baseline (Day 0), Midline (Day 45), and Endline (Day 90)
  Assessment of participants' libido using a Libido Questionnaire. These assessments will be conducted at Baseline (Day 2-5 of the first menstrual period), Midline (Day 2-5 of the second menstrual period), and Endline (Day 2-5 of the third menstrual period).

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No